CLINICAL TRIAL: NCT05819359
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of BIA 28-6156 in Subjects With Parkinson's Disease With a Pathogenic Variant in the Glucocerebrosidase (GBA1) Gene
Brief Title: Efficacy, Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of BIA 28-6156 in GBA-PD
Acronym: ACTIVATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bial R&D Investments, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA 28-6156-201; 2022-501783-18-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson Disease; Neurodegenerative Diseases; Central Nervous System Diseases; Glucocerebrosidase (GCase) activity; Parkinsonian Disorders; Basal Ganglia Diseases; Movement Disorders; GBA1 gene; BIA 28-6156; Phase 2
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Central Nervous System Diseases; Motor Activity; Parkinsonian Disorders; Basal Ganglia Diseases; Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BIA 28-6156 10 mg (Experimental): Participants will be randomized to receive BIA 28-6156 10 mg during the Treatment Period.
  Interventions: Drug: BIA 28-6156 10 mg
- BIA 28-6156 60 mg (Experimental): Participants will be randomized to receive BIA 28-6156 60 mg during the Treatment Period.
  Interventions: Drug: BIA 28-6156 60 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIA 28-6156 10 mg — BIA 28-6156 10 mg, once daily, oral administration.
  Arms: BIA 28-6156 10 mg
Drug: BIA 28-6156 60 mg — BIA 28-6156 60 mg, once daily, oral administration.
  Arms: BIA 28-6156 60 mg
Drug: Placebo — Placebo, once daily, oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled study is to assess the efficacy of BIA 28-6156 over placebo in delaying clinical meaningful motor progression over 78 weeks in subjects with Parkinson's disease who have a pathogenic variant in the glucocerebrosidase 1 (GBA1) gene (GBA-PD).

DETAILED DESCRIPTION:
This is a 2-part (Part A [Genetic Screening] and Part B [Double-Blind Treatment]), Phase 2, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, tolerability, pharmacodynamics, and pharmacokinetics of 2 fixed dose levels of BIA 28-6156 (10 and 60 mg/day) in approximately 237 subjects with genetically confirmed GBA-PD.

Part A (Genetic Screening) will identify individuals with a PD risk-associated variant in the GBA1 gene for potential enrolment into Part B (Double-Blind Treatment) of the study. Part B will consist of a screening period to ensure that all protocol inclusion/exclusion criteria for Part B of the study are met (up to 5 weeks). After screening period, eligible subjects will be randomized into 1 of 3 treatment arms (BIA 28-6156 10 mg/day, BIA 28-6156 60 mg/day, or placebo) in a 1:1:1 ratio, and enter a double-blind treatment period up to 78 weeks, followed by a 30-day (4 weeks) of safety follow-up period.

Subjects must be receiving a stable dose of PD medication for at least 30 days before screening (for Part B [Double-Blind Treatment]) and will continue to receive their usual PD medications throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects who satisfy all of the following criteria will be eligible for Part A (Genetic Screening) of the study:

* The subject is ≥35 and ≤80 years of age at the time of informed consent.
* The subject has a clinical diagnosis of PD for at least 1 year and for no longer than 7 years before initiation of screening (for Part A), as confirmed by a neurologist using the MDS Criteria for Parkinson's Disease.
* The subject has a modified Hoehn and Yahr score ≤2.5.
* The subject is receiving symptomatic treatment for PD.
* The subject is capable of giving signed informed consent.

Subjects who satisfy all the following criteria will be eligible for Part B (Double-Blind Treatment) of the study:

* Informed Consent - The subject is capable of giving signed informed consent.
* The subject has a known GBA-PD risk-associated variant (as determined in Part A [Genetic Screening] of this study).
* The subject has a score ≥22 on the Montreal Cognitive Assessment (MoCA) scale.
* The subject does not have severe motor fluctuations or disabling dyskinesias in the clinical judgment of the investigator.
* The subject has been on stable doses of PD medications for at least 30 days (at least 60 days for rasagiline) before initiation of screening in Part B (Double-Blind Treatment).
* The subject is able to comply with the study restrictions.
* The subject has a body mass index (BMI) of 18 to 40 kg/m2.
* If a sexually active man or a women of childbearing potential, the subject agrees to use highly effective birth control or to remain abstinent during the trial and for 30 days after the last dose of IMP. Complete abstinence from sexual intercourse if this is the subject's usual and preferred lifestyle; or sexual partner with surgical sterilization (e.g., tubal ligation, hysterectomy and/or bilateral oophorectomy, vasectomy).

Exclusion Criteria:

• Individuals who do not satisfy the inclusion criteria for Part A (Genetic Screening) will be excluded.

Subjects who meet any of the following criteria for Part B (Double-Blind Treatment) are not eligible for the study.

* The subject has Gaucher's disease (GD), as defined by clinical signs and symptoms (i.e., hepatosplenomegaly, cytopenia, skeletal disease), and/or a medical history of marked deficiency of GCase activity compatible with GD.
* The subject is homozygous for a GBA1 pathogenic variant that is known to be associated with GD or compound heterozygous for 2 alleles that are known to be associated with GD.
* The subject carries a known PD-associated LRRK2 pathogenic variant.
* The subject has atypical or secondary parkinsonism by medical history or in the opinion of the investigator. Atypical parkinsonism includes, but is not limited to, diagnoses of progressive supranuclear palsy, cortico-basal syndrome, and multiple system atrophy. Secondary parkinsonism includes drug-induced, toxin-induced, postinfectious, posttraumatic, or vascular parkinsonism.
* The subject has a history of (within 60 days before initiation of screening) or has planned upcoming major surgery that could interfere with, or for which the treatment might interfere with, the conduct of the study or that would pose an unacceptable risk to the subject in the opinion of the investigator.
* The subject has any active or chronic disease or condition other than PD that could interfere with, or for which the treatment might interfere with, the conduct of the study or pose an unacceptable risk to the subject in the opinion of the investigator based on medical history, physical examination, vital signs, 12-lead ECG, or clinical laboratory tests. Minor deviations of laboratory values from the normal range may be acceptable if judged by the investigator to have no/minor clinical relevance.
* The subject has a recent history (last 6 months) of abuse of addictive substances (alcohol, illegal substances), currently uses >21 units of alcohol per week, or is a regular recreational user of sedatives, hypnotics, tranquillizers, or any other addictive agent in the opinion of the investigator.
* The subject has a positive test for drugs of abuse at screening or before administration of the first dose of investigational medicinal product (IMP) that the investigator judges as clinically relevant. A positive test for tetrahydrocannabinol (THC) is exclusionary. A positive test for cannabinoids (not containing THC) is not exclusionary if the subject is a recreational user (not an abuser) of cannabinoids, in the opinion of the investigator, and agrees to abstain from using cannabinoids within 12 hours before study visits. A positive drug screen that is attributed to an allowed prescription drug is not exclusionary but should be agreed with the medical monitor.
* The subject is currently pregnant, is planning pregnancy within the timeframe of the study, or is breastfeeding.
* The subject is using a strong inhibitors and inducers CYP3A4 at the time of screening for Part B (Double-Blind Treatment).
* The subject is using a breast cancer resistance protein (BCRP) substrate (e.g., pravastatin, rosuvastatin, glyburide) at the time of screening for Part B (Double-Blind Treatment).
* The subject has used any of the following medications within 60 days before Baseline: typical or atypical antipsychotics (including, but not limited to, clozapine, pimavanserin, olanzapine, risperidone, and aripiprazole), metoclopramide, prochlorperazine, methyldopa, tetrabenazine, deutetrabenazine, valbenazine, or reserpine.
* The subject has received a vaccination within 14 days before administration of the first dose of IMP.
* The subject has a prior history of or there is a plan to conduct deep brain stimulation (DBS), lesional procedures, (i.e., thalamotomy), or focused ultrasound; to initiate gene therapy treatment for PD; or to initiate use of any formulation of intestinal infusion or continuous subcutaneous infusion of PD medications.
* The subject is currently participating in or has participated in an investigational drug study within 3 months or 5 half-lives, whichever is longer; in a therapeutic device study within 3 months before the first dose of IMP; or has previously participated in a gene therapy trial. Concurrent participation in an observational study is acceptable.
* The subject has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV), or human immunodeficiency virus 1 (HIV-1) or 2 (HIV-2) at screening. If reflex testing for hepatitis B or HCV DNA is negative, the subject may be eligible for the study.
* The subject has renal insufficiency as defined by an estimated glomerular filtration rate (eGFR) of <60 mL/min at screening.
* The subject has cirrhosis (Child-Pugh A, B, or C) or any of the following laboratory values at screening: serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN) or bilirubin >2 × ULN except if the subject has known or suspected Gilbert's disease.
* The subject has a QT interval corrected for heart rate by Fridericia's method (QTcF) value >450 msec if male or >470 msec if female at screening.
* The subject provides a positive response on Question 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) based on the last 6 months or, in the opinion of the investigator, presents a serious risk of suicide at screening.
* The subject had a positive severe acute respiratory syndrome-related coronavirus-2 (SARS-CoV-2) test (any type) result within the 30 days before signing informed consent for Part B (Double-Blind Treatment) or has 2 or more current symptoms (e.g., sore throat, cough, fever) at the same time that are consistent with the Coronavirus disease 2019 (COVID-19) infection (not tested) in the opinion of the investigator.
* The subject has a clinical history that is consistent with a previous COVID-19 infection and has not recovered fully, maintaining nonspecific symptoms like, for example, fatigue, shortness of breath, difficulty concentrating, sleep disorders, fever, anxiety, and depression.
* The subject has previously received BIA 28-6156 or has a known allergy or hypersensitivity to BIA 28-6156 or any components of the formulation.
* The subject is an unsuitable candidate to receive BIA 28-6156 or is unable or unlikely to comply with the dosing schedule or study evaluations in the judgment of the investigator.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Time from baseline to clinically meaningful progression on motor aspects of experiences of daily living (assessed by MDS-UPDRS Part II score and MDS-UPDRS Part III score) | From Baseline up to Week 78
  Time from baseline to clinically meaningful progression on motor aspects of experiences of daily living, as assessed by ≥2-point increase from baseline in Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II score and no improvement in the Motor Examination, as assessed by ≥0-point increase from baseline in MDS-UPDRS Part III score. MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part II assesses motor experiences of daily living (Range 0-52). It contains 13 questions which are to be rated by the patient and/or caregiver. Part III assesses the motor signs of PD and is rated by the investigator (Range 0-132). Part III contains 33 scores based on 18 items. For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicates more severe symptoms of PD.

SECONDARY OUTCOMES:
Time from baseline to clinically meaningful progression on motor signs of the disease (assessed by MDS-UPDRS Part III score) | From Baseline up to Week 78
  Time from baseline to clinically meaningful progression on motor signs of the disease, as assessed by a ≥5-point increase from baseline in the MDS-UPDRS Part III score. MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part III assesses the motor signs of PD and is rated by the investigator (Range 0-132). Part III contains 33 scores based on 18 items. A higher score indicates more severe symptoms of PD.
Time from baseline to any worsening on the Clinical Global Impression - Change (CGI-C) scale | From Baseline up to Week 78
  The Clinical Global Impression of Change (CGI-C) is a scale used to assess the overall clinical improvement or worsening of a patient's condition over time. The CGI-C scale ranges from 1 to 7, with lower scores indicating greater improvement (1 - Very much improved, 2 - Much improved, 3 - Minimally improved, 4 - No change, 5 - Minimally worse, 6 - Much worse, 7 - Very much worse).
Time from baseline to any worsening on the Patient Global Impression - Change (PGI-C) scale | From Baseline up to Week 78
  The Patient Global Impression of Change (PGI-C) is a self-report tool used to assess a patient's perception of their overall improvement or worsening in a particular health-related domain over time. The PGI-C scale asks patients to rate their overall improvement or worsening since the start of treatment on a seven-point scale, with lower scores indicating greater improvement (1 - Very much improved, 2 - Much improved, 3 - Minimally improved, 4 - No change, 5 - Minimally worse, 6 - Much worse, 7 - Very much worse)
Change from Baseline to Week 78 in the MDS-UPDRS Total (Part I-IV) score | From Baseline up to Week 78
  The MDS-UPDRS assesses nonmotor and motor experiences of daily living, motor examination, and motor complication categories. The MDS-UPDRS Part I-IV total score was calculated as the sum of the individual item scores from these categories. Each item is rated on a scale from 0 to 4 on which 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. A higher score indicates more severe symptoms of PD.
Change from Baseline to Week 78 in the Modified Hoehn and Yahr score | From Baseline up to Week 78
  The Modified Hoehn and Yahr scale measures the severity of Parkinson's disease by assessing the patient's motor symptoms and functional impairment. The scale has seven stages, ranging from 1 to 5, with higher scores indicating more severe disease. (1 - Unilateral involvement only; 1.5 - Unilateral and axial involvement; 2 - Bilateral involvement without impairment of balance; 2.5 - Mild bilateral disease with recovery on pull test; 3 - Mild to moderate bilateral disease; some postural instability; physically independent; 4 - Severe disability; still able to walk or stand unassisted; 5 - Wheelchair bound or bedridden unless added).
Change from Baseline to Week 78 in the 39-Item Parkinson's Disease Questionnaire (PDQ-39) score | From Baseline up to Week 78
  The PDQ-39 is the most thoroughly validated and extensively used self-report measure for the assessment of health-related quality of life in patients with PD. The questionnaire measures 39 items, which assess 8 domains of health: mobility (10 items), activities of daily living (6 items), emotional well being (6 items), stigma (4 items), social support (3 items), cognitions (4 items), communication (3 items), and bodily discomfort (3 items). Each item is scored on the following scale: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, and 4 = always. Items in each subscale and the total scale can be summarized into an index and transformed linearly to a scale from 0 (perfect health as assessed by the measure) to 100 (worst health as assessed by the measure).

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Costa, Study Director — Bial R&D Investments, S.A.
Locations (95):
- United States (43):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - Cedars-Sinai, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Parkinson's Center and Movement Disorders of Boca Raton, Boca Raton, Florida
  - University of Miami, Dept. of Neurology, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Baylor University Medical Center, Baltimore, Maryland
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Quest Research Institute, LLC, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Struthers Parkinson's Center- East, Saint Paul, Minnesota
  - Park Nicollet Struther's Parkinson's Center (Struthers Parkinsons Center at HealthPartners), Saint Paul, Minnesota
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai Beth Israel, New York, New York
  - Weil Cornell Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Northwell Health Physician Partners, New York, New York
  - Northwell Health, New York, New York
  - University of Rochester Neurology, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, South Euclid, Ohio
  - Univerity of Toledo, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Parkinson's Disease and Movement Disorders Cente at University of Pennyslvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center - San Antonio, San Antonio, Texas
  - Intermountain Healthcare, Salt Lake City, Utah
  - Evergreen Neuroscience Institute, Kirkland, Washington
  - University of Washington, Seattle, Washington
  - Inland Northwest Research, Spokane, Washington
- Canada (3):
  - Clinique Neuro-Outaouais (Neuro-Outaouais Clinic), Gatineau, Quebec
  - Montreal Neurological Institute & Hospital, Montreal, Quebec
  - Ottawa Hospital Research Institute, Ottawa
- France (7):
  - CHU de Nantes - Hopital Nord Laennec, Nantes
  - CHU de Nice Hopital Pasteur, Nice
  - CHU de Nimes, Nîmes
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Pitie-Salpetriere - Centres d'Investigation Clinique (CIC) Paris-Est, Paris
  - CHU de Rennes Hopital Pontchaillou, Rennes
  - CIC Toulouse, Toulouse
  - Hopital Paule de Viguier, Toulouse
- Germany (7):
  - Neurologisches Fachkrankenhaus für, Bewegungsstörungen und Parkinson, Beelitz-Heilstätten
  - Gertrudis Clinic Biskirchen, Parkinson-Center, Biskirchen
  - Paracelsus-Elena-Klinik, Kassel
  - Universitats klinikum Marburg, Marburg
  - Klinikum der Universität München, Campus Grosshadern, Neurologische Klinik und Poliklinik, Munich
  - Ludwig-Maximilians University Munich, Munich
  - Parkinson-Klinik Ortenau GmbH&Co KG, Wolfach
- Italy (10):
  - IRCCS Istituto Delle Scienze Neurologiche DI, Bologna
  - Spedali Civilia di Brescia, Brescia
  - Ospedale Antonio Perrino, Brindisi
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Carlo Besta Neurological Institute, Milan
  - Universita degli Studi della Campania Luigi Vanvitelli - Clinica Neurologia I, Napoli
  - Universita degli Studi di Padova - Azienda Ospedaliera di Padova - Clinica Neurologica, Padua
  - IRCSS San Raffaele Pisana, Roma
  - Istituto Clinico Humanitas, Rozzano
  - A.O.U. San Giovanni di Dio Ruggi d'Aragona Centro Parkinson- Piano Rialzato Corpo QT, Salerno
- Netherlands (3):
  - Amsterdam Medical Center UMC, Amsterdam
  - University Medical Center Groningen, Groningen
  - St. Antonius Ziekenhuis (St. Antonius Hospital) - Utrecht, Utrecht
- Poland (3):
  - Centrum Medyczne NEUROMED Sp. z o.o. ul., Bydgoszcz
  - Krakowkska Akademia Neurologii Sp. z o.o, Krakow
  - NeuroKlinika Gabinet Lekarski, Lodz
- Portugal (5):
  - Centro Hospitalar Universitario de Coimbra, Coimbra
  - Hospital Senhora da Oliveira de Guimaraes, Guimarães
  - Centro Hospitalar Universitario de Santo Antonio, Porto
  - Hospital S.JOÃO, Porto
  - CNS - Campus Neurologico, Torres Vedras
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitario Cruces, Barakaldo
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Vall D´Hebron, Barcelona
  - Hospital Universitaio de La Princesa, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Sweden (2):
  - Skane University Hospital, Lund University, Lund
  - Neurologmottagningen, QD 62, Uppsala
- United Kingdom (5):
  - NHS Tayside-Ninewells Hospital and Medical School, Dundee
  - Glasgow Memory Clinic, Glasgow
  - King's College London - David Goldberg Centre, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Freeman Hospital, Newcastle upon Tyne
  - University Hospitals Plymouth NHS Trust, Plymouth